CLINICAL TRIAL: NCT01071915
Title: An Open-label, Multi-Centre Trial, Bridging Efficacy and Safety of Degarelix One-Month Dosing Regimen in Korean Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Brief Title: Efficacy and Safety of Degarelix One Month Dosing Regimen in Korean Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Pharmaceuticals Korea, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS42
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix 240/80 mg (Experimental): The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The subsequent maintenace of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections at 28 day intervals from day 28 to day 168.
  Interventions: Drug: Degarelix 240/80 mg

INTERVENTIONS:
Drug: Degarelix 240/80 mg — The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The subsequent maintenance doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections at 28 day intervals from day 28 to day 168.
  Other Names: FE200486; FIRMAGON

SUMMARY:
This is an open-label, multi-centre single arm trial to investigate efficacy and safety of degarelix in Korean patients with prostate cancer for bridging between CS21 trial (NCT00295750) results.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent before any trial-related activity is performed.
* Has a histologically confirmed (Gleason graded) adenocarcinoma of the prostate (all stages) (except for neoadjuvant hormonal therapy/ includes patients with rising PSA after prostatectomy or radiotherapy)
* Is a male patient aged 18 years or older
* Has a screening serum testosterone level >1.5 ng/mL
* Has an ECOG (Eastern Cooperative Oncology Group) score of ≤ 2
* Has a screening PSA value of ≥2 ng/mL
* Has a life expectancy of at least 12 months

Exclusion Criteria:

* Has had previous or is currently under hormonal management of prostate cancer. However, prostatectomy or radiotherapy with curative intention, neoadjuvant/adjuvant hormonal therapy are accepted for a maximum duration of 6 months, at least 6 months prior to Screening Visit
* Is currently treated with a 5-α-reductase inhibitor
* Is considered to be candidate for curative therapy, i.e. radical prostatectomy or radiotherapy
* Has a history of severe untreated asthma, anaphylactic reactions or severe urticaria and/or angioedema
* Has hypersensitivity towards any component of the investigational medicinal product
* A marked baseline prolongation of QT/QTcF interval
* A history of additional risk factors for Torsade de Pointes ventricular arrhythmias
* Has had cancer within the last five years except prostate cancer and surgically removed basal or squamous cell carcinoma of the skin
* Has a known or suspect hepatic, symptomatic biliary disease
* Has elevated serum ALT level more than the upper limit of normal or serum total bilirubin level above the upper level of normal range at the Screening Visit and confirmed with a second measurement within 21 days
* Has other clinically significant laboratory abnormalities
* Has a clinically significant disorder (other than prostate cancer) or any other condition, including alcohol or drug abuse
* Has a mental incapacity or language barriers precluding adequate understanding or co- operation
* Has received an investigational drug within the last 28 days preceding Screening Visit or longer if considered to possibly influence the outcome of the current trial
* Has previously participated in any degarelix trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (11):
- South Korea (11):
  - Kyoungbuk National University Hospital, Daegu, Daegu
  - Hallym University Sacred Heart Hospital, Pyungchon, Gyunggi-do
  - Pusan National University Yangsan Hospital, Mulgeum-eup, Gyungnam
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Yonsei University Health System (Sevrance Hospital), Seoul
  - Yonsei University Health System Gangnam Sevrance, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from 11 sites in Korea. The study was conducted between 08 March 2010 (FPFV) and 07 November 2011 (LPLV).
Period: Overall Study
Arm/Group | Degarelix 240/80 mg
Started | 157 (Intention to Treat Analysis Set)
Full Analysis Set (FAS) | 155
Safety Analysis Set | 156
Completed | 148
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — Miscellaneous Reasons | 2

BASELINE CHARACTERISTICS:
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 155
Age Continuous [Mean (Standard Deviation); unit: years] | 72.6 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline values based on FAS
  Participants
    Female | 0
    Male | 155
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 155
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 23.8 (2.98)
Gleason Score [Number; unit: Participants] — FAS. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  1 patient did not have a Gleason Score
  Participants
    Gleason Score 2-4 | 0
    Gleason Score 5-6 | 24
    Gleason Score 7-10 | 130
Stage of Prostate Cancer [Number; unit: Participants] — FAS. Prostate cancer stage was classified according to the Tumor, Nodes, and Metastatic (TNM) scale to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor. Some participants did not have their prostate cancer classified for the complete TNM scale (13 participants).
  Participants
    Localized | 43
    Locally Advanced | 60
    Metastatic | 39
    Not Classifiable | 13
Serum Testosterone Level [Median (Full Range); unit: nanograms per milliliter (ng/mL)] | 4.03 [1.08 to 10.7]
Serum Protsate-Specific Antigen (PSA) Levels [Median (Full Range); unit: ng/mL] | 19.2 [1.59 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Probability of Testosterone at Castrate Level (≤0.5 ng/mL) From Day 28 to Day 196
Time Frame: Day 28 to Day 196
Population: 152 participants for this outcome measure is the analysis population from day 28 to day 196
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 152
percent probability | 96.7 [92.2 to 98.6]

2. Secondary Outcome: Proportion of Patients With Testosterone Level ≤0.5 ng/mL at Day 3
Time Frame: At day 3
Population: Observed cases
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 154
percent | 97.4 [93.5 to 99.3]

3. Secondary Outcome: Percentage Change in Prostate-specific Antigen (PSA) From Baseline to Day 28
Time Frame: To Day 28
Population: 152 participants for this outcome measure is the analysis population from day 0 to day 28
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 152
percent | -79.7 [-90.5 to -64.5]

4. Secondary Outcome: Cumulative Probability of Testosterone at Castrate Level (≤0.5 ng/mL)From Day 56 to Day 196
Time Frame: Day 56 to Day 196
Population: 152 participants for this outcome measure is the analysis population from day 56 to day 196
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 152
percent probability | 96.7 [92.2 to 98.6]

5. Secondary Outcome: Cumulative Probability of no PSA Failure From Day 28 to Day 196
Description: PSA failure was defined as two consecutive increases of 50%, and at least 5 ng/mL, compared to nadir.
Time Frame: To Day 196
Population: 152 participants for this outcome measure is the analysis population from day 28 to day 196
Measure: Mean (95% Confidence Interval); unit: percent probability
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 152
percent probability | 97.3 [93.1 to 99.0]

6. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables
Description: The figures present the number of participants who had markedly abnormal levels of safety laboratory variables. Only the laboratory variables that had at least one percentage of participants in either group with abnormal value are presented, more variables were included in the study.
Time Frame: To Day 196
Population: Safety analysis population
Measure: Number; unit: participants
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 156
participants
  B-Haematocrit (Ratio) <=0.37 | 73
  B-Haemoglobin (g/L) <=115 | 5
  B-White blood cell count (10^9/L) <=2.8 | 1
  B-White blood cell count (10^9/L) >=16.0 | 1
  B-Red blood cell count (10^12/L) <=3.5 | 19
  S-Alanine aminotransferase (IU/L) >3xULN | 1
  S-Potassium (mmol/L) >=5.8 | 10
  S-Sodium (mmol/L) <=130 | 2
  S-Urea nitrogen (mmol/L) >=10.7 | 8
  B-Lymphocytes (%) <=10 | 4
  B-Eosinophils (%) >=10 | 7

7. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: To Day 196
Population: Safety analyis population
Measure: Number; unit: participants
Arm/Group | Degarelix 240/80 mg
Number analyzed (Participants) | 156
participants
  Diastolic blood pressure <=50 and decrease >=15 | 6
  Diastolic blood pressure >=105 and increase >=15 | 0
  Systolic blood pressure <=90 and decrease >=20 | 12
  Systolic blood pressure >=180 and increase >=20 | 1
  Heart rate <=50 and decrease >=15 | 4
  Heart rate >=120 and increase >=15 | 0
  Body weight decrease of >=7 percent | 4
  Body weight increase of >=7 percent | 12

ADVERSE EVENTS:
Time Frame: 7 months (196 days)
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix 240/80 mg
Serious Adverse Events (participants affected / at risk) | 18/156
Other Adverse Events (participants affected / at risk) | 113/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 240/80 mg (N=156)
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Disease progression (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraplegia (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Ureteral stent removal (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 240/80 mg (N=156)
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 5
Injection site pain (General disorders) | 34
Injection site erythema (General disorders) | 13
Injection site induration (General disorders) | 6
Oedema peripheral (General disorders) | 6
Fatigue (General disorders) | 5
Upper respiratory tract (Infections and infestations) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 6
Insomnia (Nervous system disorders) | 7
Nocturia (Renal and urinary disorders) | 10
Dysuria (Renal and urinary disorders) | 6
Haematuria (Renal and urinary disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14
Hot flush (Vascular disorders) | 5
Flushing (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.